CLINICAL TRIAL: NCT02614898
Title: Evidence - Evaluation of Potential Predictors of Disease Progression in Patients With aHUS, Including Genetics, Biomarkers and Treatment
Brief Title: Evaluation of Potential Predictors of Disease Progression in Participants With Atypical Hemolytic Uremic Syndrome (aHUS) Including Genetics, Biomarkers, and Treatment
Acronym: EVIDENCE
Status: Terminated | Type: Observational
Why Stopped: Terminated for administrative reasons before enrollment was complete.
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ECU-aHUS-403; 2015-003135-35 (EudraCT Number)
Record Dates: First submitted 2015-11-24; First posted 2015-11-25 (Estimated); Results first posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Atypical Hemolytic Uremic Syndrome
MeSH Terms: conditions — Atypical Hemolytic Uremic Syndrome | interventions — eculizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Eculizumab: The targeted population consists of pediatric and adult participants with aHUS who received eculizumab at the discretion of the treating physician.
  Interventions: Other: Eculizumab

INTERVENTIONS:
Other: Eculizumab — This study was an observational study. Therefore, the study drug was not provided as part of this study, and the dosing regimen was based solely at the discretion of the treating physician.
  Other Names: Soliris®

SUMMARY:
This was a prospective, open-label study with no participant randomization. Treatment for aHUS was observational and at the discretion of the treating physician. The purpose of this study was to assess disease manifestations of complement-mediated thrombotic microangiopathy (TMA) and evaluate potential clinical predictors of disease manifestations and progression in participants with aHUS with or without eculizumab treatment in the clinical setting.

ELIGIBILITY:
Inclusion Criteria:

1. Currently receiving eculizumab treatment in the M11-001 aHUS Registry
2. Two normal platelet counts at least 4 weeks apart
3. Two normal lactate dehydrogenase levels at least 4 weeks apart
4. Willing, committed, and able to return for all clinic visits and complete all study-related procedures
5. Participant or participant's parent/legal guardian must have been willing and able to give written informed consent. Participant (if minor) must have been willing to give written informed assent (if applicable as determined by the central Institutional Review Boards/Independent Ethics Committees)

Exclusion Criteria:

1. Any prior eculizumab treatment discontinuation
2. On chronic dialysis (defined as ≥3 months on dialysis)
3. Currently participating in another complement inhibitor trial
4. Life expectancy of <6 months
5. Participant or participant's parent/legal guardian was unable to give written informed consent. Participant (if minor) was unable to give written informed assent (if applicable as determined by the central Institutional Review Boards/Independent Ethics Committees)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with aHUS enrolled in the M11-001 aHUS Registry and currently receiving eculizumab with no prior intentional eculizumab discontinuations at any time (for example, not occasional, unplanned, or temporary missed doses of eculizumab, but intended long-term discontinuation).
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2015-11-04 (Actual); Primary Completion 2017-10-05 (Actual); Study Completion 2017-10-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (8):
  - Clinical Trial Site, Washington D.C., District of Columbia
  - Clinical Trial Site, Atlanta, Georgia
  - Clinical Trial Site, Chicago, Illinois
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Hackensack, New Jersey
  - Clinical Trial Site, Charlotte, North Carolina
  - Clinical Trial Site, Columbus, Ohio
  - Clinical Trial Site, Houston, Texas
- Australia (10):
  - Clinical Trial Site, Adelaide
  - Clinical Trial Site, Clayton
  - Clinical Trial Site, Heidelberg
  - Clinical Trial Site, Kingswood
  - Clinical Trial Site, Liverpool
  - Clinical Trial Site, Nedlands
  - Clinical Trial Site, Parkville
  - Clinical Trial Site, Perth
  - Clinical Trial Site, Westmead
  - Clinical Trial Site, Woolloongabba
- Germany (4):
  - Clinical Trial Site, Hannover
  - Clinical Trial Site, Hanover
  - Clinical Trial Site, Kiel
  - Clinical Trial Site, Lübeck
- Clinical Trial Site, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Sixty-seven participants were enrolled in this study (15 pediatric and 52 adults). Treatment information was missing for 1 adult participant.
Groups:
- Pediatric: Participants with atypical hemolytic uremic syndrome (aHUS) who were less than 18 years at baseline and who initiated treatment with eculizumab prior to study entry. Dosing regimen changed solely at the discretion of the treating physician.
- Adult: Participants with aHUS who were 18 years or older at baseline and who initiated treatment with eculizumab prior to study entry. Dosing regimen changed solely at the discretion of the treating physician.
Period: Overall Study
Arm/Group | Pediatric | Adult
Started | 15 | 52
Safety Population | 15 | 52
Completed | 0 | 1
Not Completed | 15 | 51
Not completed — Participated until study termination | 10 | 26
Not completed — Lost to Follow-up | 0 | 2
Not completed — Physician Decision | 1 | 8
Not completed — Study Terminated by Sponsor | 3 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Withdrawal by Parent/Guardian | 1 | 1
Not completed — Other-Additional Information Unavailable | 0 | 11
Not completed — Missing | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Pediatric: Participants with aHUS who were less than 18 years at baseline and who initiated treatment with eculizumab prior to study entry. Dosing regimen changed solely at the discretion of the treating physician.
- Total: Total of all reporting groups
Arm/Group | Pediatric | Adult | Total
Number analyzed (Participants) | 15 | 52 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.9 (3.46) | 43.3 (17.26) | 35.4 (21.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 34 | 40
  Male | 9 | 18 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 12 | 44 | 56
  Asian | 1 | 2 | 3
  Black | 1 | 5 | 6
  Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Rate Of Thrombotic Microangiopathy (TMA) Manifestations During Eculizumab Treatment Compared To Off-Treatment
Description: A TMA manifestation was defined as one of following: Hematologic or renal events due to aHUS; extra-renal clinical signs and symptoms of aHUS; tissue (for example, kidney transplant) biopsy demonstrating TMA due to aHUS.
  The study was terminated with only 20% of the planned enrollment and due to the subsequent loss of funding for the program, the samples collected for outcome measure assessment could not be analyzed to generate summary-level data. All participants enrolled in ECU-aHUS-403 were concurrently enrolled in protocol M11-001, and their data will be included in the analyses for M11-001.
Time Frame: Baseline, 24 Months
Population: All enrolled participants. The study was terminated with only 20% of the planned enrollment; because the program lost funding, samples collected could not be analyzed to generate summary-level data. All participants enrolled in ECU-aHUS-403 were concurrently enrolled in protocol M11-001, and their data will be included in the analyses for M11-001.
Arm/Group | Pediatric | Adult
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change From Baseline To 24 Months In Estimated Glomerular Filtration Rate (eGFR)
Description: Change in estimated eGFR over time using the chronic kidney disease-epidemiology (CKD-EPI) formula.
  The study was terminated with only 20% of the planned enrollment and due to the subsequent loss of funding for the program, the samples collected for outcome measure assessment could not be analyzed to generate summary-level data. All participants enrolled in ECU-aHUS-403 were concurrently enrolled in protocol M11-001, and their data will be included in the analyses for M11-001.
Time Frame: Baseline, 24 Months
Population: as for outcome 1
Arm/Group | Pediatric | Adult
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Incidence Of Plasma Exchange And Plasma Infusion (PE/PI)
Description: The number of occurrences of PE/PI per participant-years was calculated and summarized by treatment status.
  The study was terminated with only 20% of the planned enrollment and due to the subsequent loss of funding for the program, the samples collected for outcome measure assessment could not be analyzed to generate summary-level data. All participants enrolled in ECU-aHUS-403 were concurrently enrolled in protocol M11-001, and their data will be included in the analyses for M11-001.
Time Frame: Baseline, 24 Months
Population: as for outcome 1
Groups:
- Adult: Participants with aHUS who were 18 years or older at baseline and who were treated with eculizumab. Dosing regimen changed solely at the discretion of the treating physician.
Arm/Group | Pediatric | Adult
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 0 through Month 24
Arm/Group | Pediatric | Adult
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/52
Serious Adverse Events (participants affected / at risk) | 1/15 | 14/52
Other Adverse Events (participants affected / at risk) | 6/15 | 31/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pediatric (N=15) | Adult (N=52)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 1
Liver injury (Hepatobiliary disorders) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Cellulitis streptococcal (Infections and infestations) | 0 | 1
Cytomegalovirus viraemia (Infections and infestations) | 0 | 1
Device related sepsis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 2
Influenza (Infections and infestations) | 1 | 0
Metapneumovirus infection (Infections and infestations) | 1 | 0
Rhinovirus infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 2
Hemiparesis (Nervous system disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Drug abuse (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 2
Acute lung injury (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Pediatric (N=15) | Adult (N=52)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 1
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Bradycardia (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 1
Inner ear inflammation (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Blindness unilateral (Eye disorders) | 0 | 1
Eye colour change (Eye disorders) | 0 | 1
Eye disorder (Eye disorders) | 0 | 1
Ocular icterus (Eye disorders) | 0 | 1
Orbital oedema (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 6
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1
Anal incontinence (Gastrointestinal disorders) | 0 | 1
Anorectal discomfort (Gastrointestinal disorders) | 0 | 1
Bowel movement irregularity (Gastrointestinal disorders) | 0 | 1
Chronic gastritis (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 7
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastrointestinal erosion (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Malabsorption (Gastrointestinal disorders) | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 11
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 4
Asthenia (General disorders) | 0 | 7
Catheter site erythema (General disorders) | 0 | 1
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 2
Extravasation (General disorders) | 0 | 1
Face oedema (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 6
Feeling hot (General disorders) | 0 | 1
Hypothermia (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 2
Peripheral swelling (General disorders) | 0 | 3
Pyrexia (General disorders) | 1 | 3
Temperature intolerance (General disorders) | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1
Aeromonas infection (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Catheter site infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 2
Escherichia urinary tract infection (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 3
Oral herpes (Infections and infestations) | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 2
Tonsillitis (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 11
Urinary tract infection (Infections and infestations) | 0 | 3
Varicella zoster virus infection (Infections and infestations) | 0 | 1
Viral pharyngitis (Infections and infestations) | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0/6 | 2/34
Anal injury (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Corneal abrasion (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Procedural dizziness (Injury, poisoning and procedural complications) | 1 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1
Blood calcium increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 5
Blood lactate dehydrogenase increased (Investigations) | 0 | 2
Blood magnesium decreased (Investigations) | 0 | 1
Bone density decreased (Investigations) | 0 | 1
Faecal calprotectin increased (Investigations) | 0 | 1
Faecal elastase concentration decreased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Haptoglobin decreased (Investigations) | 1 | 0
Liver function test increased (Investigations) | 0 | 1
Red blood cell schistocytes present (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 3
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3
Angiolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Dizziness postural (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 10
Hypotonia (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 2
Migraine (Nervous system disorders) | 0 | 1
Poor quality sleep (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 3
Confusional state (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Irritability (Psychiatric disorders) | 0 | 5
Dysuria (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 2
Renal impairment (Renal and urinary disorders) | 0 | 1
Renal tubular acidosis (Renal and urinary disorders) | 0 | 1
Amenorrhoea (Reproductive system and breast disorders) | 0/6 | 1/34
Breast cyst (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 6
Hypotension (Vascular disorders) | 0 | 5
Thrombophlebitis (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
As the study was terminated for administrative reasons, before enrollment was complete, and the program subsequently lost funding, all collected data could not be analyzed to generate summary-level data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-05): https://cdn.clinicaltrials.gov/large-docs/98/NCT02614898/Prot_SAP_000.pdf